CLINICAL TRIAL: NCT00511381
Title: Utility of Genetic Testing in Detection of Late-Onset Hearing Loss
Brief Title: Genetic Testing in Detection of Late-Onset Hearing Loss
Acronym: SoundGene
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: PDX-001-07
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Hearing Loss; Late-Onset Hearing Loss; Deafness
Keywords: Hearing Loss; Late-Onset Hearing Loss; Deafness
MeSH Terms: conditions — Hearing Loss; Deafness

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: No intervention — No intervention

SUMMARY:
Two major limitations of existing audiometric newborn hearing screening programs are their inability to detect forms of deafness that are not expressed at birth and the low compliance with obtaining recommended audiologic confirmation and/or follow-up. Molecular genetic tests on blood spots from all newborns will identify those at risk for the most frequent causes of late-onset hearing loss and to add these infants to the group who should receive continued audiologic monitoring.

DETAILED DESCRIPTION:
Two major limitations of existing audiometric newborn hearing screening programs are their inability to detect forms of deafness that are not expressed at birth and the low compliance with obtaining recommended audiologic confirmation and/or follow-up. Molecular genetic tests on blood spots from all newborns will identify those at risk for the most frequent causes of late-onset hearing loss and to add these infants to the group who should receive continued audiologic monitoring.

The specific aims of this project are to:

* Demonstrate the utility of detecting four potentially important causes of delayed onset hearing loss by molecular tests at birth, which may be missed by current audiometric screening tests.
* Document the frequency, clinical and genetic characteristics of hearing loss associated with each condition.

Dried blood spots (DBS) on filter paper will be obtained and be used for this project with parental informed consent from 6,000 newborn infants at approximately 25 hospitals. Pediatrix Screening, a subsidiary of Pediatrix Medical Group with long experience in high throughput neonatal testing, will perform genetic testing on the samples. The four genetic and environmental forms of deafness to be studied include:

* Prenatal/congenital cytomegalovirus (CMV) infection

  -Detecting the presence of CMV viral DNA in dried blood spots.
* Connexin Deafness - GJB2 and GJB6 mutations

  - Cx26 35delG, Cx26 235delC, Cx26 167delT, Cx26 M34T, and Cx30 large deletion.(Under sublicense with Athena Diagnostics, Inc: United States Patent Numbers: 5,998,147 and 6,485,908 and patents pending)
* Pendred Syndrome - SLC26A mutations

  - L236P, 1001 +1G>A, T416P, E384G
* Mitochondrial Mutations - T961C, T961G, G951A, 961 delT+C(n)Ins, G7444A, A7445G, A7445C.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of informed consent
* Inborn
* Ability to do ABR (auditory brainstem response screen technology) screening test on all participants
* Age at enrollment less than 14 days or less than or equal to 336 hours (Birth date is day 0)
* Gestational age > = 34 0/7 weeks and above. (Late preterm infants and term infants)
* No major anomalies
* Ability to obtain blood sample prior to administration of any blood product transfusion
* Subjects' parents or legal guardian willing to provide follow-up data on their child. They will need to provide a telephone contact number and address for follow-up procedures

Exclusion Criteria:

* Older than 14 days of age or 336 hours
* Receipt of a blood product prior to the ability to obtain blood sample for genetic testing (SoundGene panel)
* Any major congenital anomalies. (chromosomal abnormalities, cyanotic congenital heart disease, gastroschisis, omphalocele, diaphragmatic hernia, or other major gastrointestinal anomalies, major neurological injury or anomaly, and multiple congenital anomalies)

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3681 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Lim, ARNP, Principal Investigator — Pediatrix; Zhili Lin, MD, PhD, Study Chair — Pediatrix Screening; Reese H Clark, MD, Study Chair — Pediatrix
Locations (3):
- United States (3):
  - Stormont-Vail HealthCare, Topeka, Kansas
  - Miami Valley Hospital, Dayton, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma